CLINICAL TRIAL: NCT05089357
Title: A Prospective, Non-interventional Study to Collect Subject and Physician Satisfaction During Long Term Treatment of Glabellar Lines With Dysport® in Subjects of Chinese Origin in Real Clinical Practice
Brief Title: Non-interventional Study, Long Term Treatment on Glabellar Lines With Dysport® in Subjects of Chinese Origin
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 05PF2009
Record Dates: First submitted 2021-09-27; First posted 2021-10-22 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-02

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AbobotulinumtoxinA: Participants with moderate to severe GL received a total dose of AbobotulinumtoxinA (Dysport®), 50 U (0.25 mL total; 10 U [0.05 mL per injection site] of study drug into 5 injection sites intramuscularly: 2 injections into each corrugator muscle and 1 injection into the procerus muscle) at Visits 1, 3, and 5.
  Interventions: Biological: AbobotulinumtoxinA

INTERVENTIONS:
Biological: AbobotulinumtoxinA — Participants received a total dose of AbobotulinumtoxinA (Dysport®), 50 U (0.25 mL total; 10 U [0.05 mL per injection site] of study drug into 5 injection sites intramuscularly.

SUMMARY:
This is a prospective, longitudinal, non-interventional, multi-center study to collect subject and physician satisfaction, and treatment experience with Dysport in real clinical practice in subjects of Chinese origin.

DETAILED DESCRIPTION:
Approximately 250 subjects are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female up to 65 years of age, and of Chinese origin.
* Moderate (grade 2) or severe (grade 3) glabellar lines at max frown.
* Prior to and independent of study, subject is seeking long term treatment of their glabellar lines.
* Prior to and independent of the study participation, physician intended to treat the subject with Dysport.
* Time and ability to complete the study and comply with instructions.
* Understands the study requirements and signed the informed consent form (ICF)

Exclusion Criteria:

* Hypersensitive to Dysport or its excipients.
* Presence of contraindications to Dysport treatment as specified in the approved leaflet in China.
* Subject is at risk for precautions, warnings, and/or contraindications to Dysport as specified in the approved leaflet in China.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult subjects up to 65 years of age with moderate to severe glabellar lines (GL)
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Song, Principal Investigator — Hangzhou Yanshuyuerong medical cosmetology clinic
Locations (1):
- Hangzhou Yanshuyuerong medical cosmetology clinic, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in China from 11 November 2021 to 24 December 2023.
Pre-assignment Details: A total of 250 participants were enrolled and received study treatment.
Groups:
- AbobotulinumtoxinA: Participants with moderate to severe Glabellar lines (GL) received a total dose of AbobotulinumtoxinA (Dysport®), 50 Units (U) (0.25 milliliter [mL] total; 10 U [0.05 mL per injection site] of study drug into 5 injection sites intramuscularly: 2 injections into each corrugator muscle and 1 injection into the procerus muscle) at Visits 1, 3, and 5.
Period: Overall Study
Arm/Group | AbobotulinumtoxinA
Started | 250
Per Protocol Set (PPS) (PPS was a subset of the Full Analysis Set (FAS) that included all participants who had evaluable primary efficacy endpoints, had overall good compliance, and had no major protocol deviations during the study.) | 204
Completed | 216
Not Completed | 34
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 6
Not completed — Medical reason | 1
Not completed — Due to completion of project, participants did not enter the follow-up window period and withdrew | 2
Not completed — Pregnancy | 2

BASELINE CHARACTERISTICS:
Population: FAS included all participants who were screened, enrolled in the study, and treated at least once with study drug.
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 250
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han (East Asian) | 229
  Other | 21
Region of Enrollment [Count of Participants; unit: Participants]
  China | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Each Response Category for Overall Participant Satisfaction at Visit 6, Assessed by the Subject Satisfaction Questionnaire
Description: The participant's satisfaction with the treatment was assessed using a subject satisfaction questionnaire. At Visit 6 (that is., three weeks, after the 3rd injection) participants were asked "What is your overall satisfaction after three treatment cycles with Dysport?" Participant's response options were noted as: Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Percentage of participants in each response category were reported here.
Time Frame: Month 14
Population: PPS was a subset of the FAS that included all participants who had evaluable primary efficacy endpoints, had overall good compliance, and had no major protocol deviations during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 204
percentage of participants
  Very Satisfied | 71.1 [64.3 to 77.2]
  Satisfied | 28.9 [22.8 to 35.7]
  Dissatisfied | 0 [NA to NA] — 95 percent (%) confidence interval could not be calculated due to an insufficient number of participants with events.
  Very Dissatisfied | 0 [NA to NA] — 95 percent (%) confidence interval could not be calculated due to an insufficient number of participants with events.

2. Secondary Outcome: Percentage of Participants in Each Response Category for Overall Physician Satisfaction at Visit 6, Assessed by the Physician Satisfaction Questionnaire
Description: The physician's satisfaction with the treatment was assessed using a physician satisfaction questionnaire. At Visit 6 (i.e., three weeks, after the 3rd injection) Physician were asked "What is your overall satisfaction after three treatment cycles with Dysport?" Physician response options were noted as: Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Percentage of participants in each response category for overall physician satisfaction were reported here. Physicians were not considered enrolled but did contribute to this assessment.
Time Frame: Month 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- AbobotulinumtoxinA: Participants with moderate to severe GL received AbobotulinumtoxinA (Dysport®), total dose of 50 U (0.25 mL total; 10 U [0.05 mL per injection site] of study drug into each of the 5 injection sites) at Visits 1, 3, and 5.
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 204
percentage of participants
  Very Satisfied | 68.1
  Satisfied | 31.4
  Dissatisfied | 0.5
  Very Dissatisfied | 0

3. Secondary Outcome: Percentage of Participants Satisfied With the Treatment Assessed Using a Subject Satisfaction Questionnaire
Description: The participant's satisfaction with the treatment was assessed using a subject satisfaction questionnaire. Participants were asked "How satisfied with the aesthetic outcome in the Injected area after treatment" and "How satisfied were you with the comfort of the injection" Participant's response options were noted as: Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Percentage of participants in each response category were reported here.
Time Frame: Month 20
Population: PPS was a subset of the FAS that included all participants who had evaluable primary efficacy endpoints, had overall good compliance, and had no major protocol deviations during the study. Here" overall number of participants analyzed signified" participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 200
percentage of participants
  How satisfied are you with aesthetic outcome in injected area after treatment: Very satisfied | 53.0
  How satisfied are you with aesthetic outcome in injected area after treatment:Satisfied | 44.5
  How satisfied are you with aesthetic outcome in injected area after treatment:Dissatisfied | 2.0
  How satisfied are with aesthetic outcome in injected area after treatment:Very dissatisfied | 0.5
  How satisfied were you with comfort of injection: Very satisfied | 52.5
  How satisfied were you with comfort of injection: Satisfied | 45.5
  How satisfied were you with comfort of injection: Dissatisfied | 2.0
  How satisfied were you with comfort of injection: Very Dissatisfied | 0

ADVERSE EVENTS:
Time Frame: From start of study up to end of study (Up to 20 Months)
Description: The Safety Set included all participants who received at least 1 dose of study treatment and for whom actual data on safety endpoints were available.
Groups:
- AbobotulinumtoxinA: Participants with moderate to severe Glabellar lines (GL) received AbobotulinumtoxinA (Dysport®), total dose of 50 U (0.25 milliliter [mL] total; 10 U [0.05 mL per injection site] of study drug into each of the 5 injection sites) at Visits 1, 3, and 5.
Arm/Group | AbobotulinumtoxinA
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 1/250
Other Adverse Events (participants affected / at risk) | 107/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AbobotulinumtoxinA (N=250)
Severe leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Event was not related to the product or injection procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AbobotulinumtoxinA (N=250)
COVID-19 (Infections and infestations) | 58 — Events were not related to the product or injection procedure.
Upper respiratory tract infection (Infections and infestations) | 49 — Events were not related to the product or injection procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT05089357/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05089357/SAP_001.pdf